CLINICAL TRIAL: NCT05784909
Title: Outcomes of Water Vapor Thermal Therapy (REZUM) in Management of Symptomatic Patients With Benign Prostatic Enlargement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Zamra, specialist of urology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REZUM in Assiut
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients diagnosed with bladder outlet obstruction due to BPH (Experimental): all symptomatic patients with BPH with failure medical management or prefer minimal invasive procedure from the start.
  Interventions: Device: rezum

INTERVENTIONS:
Device: rezum — Technique With the patient in a lithotomy position, after cystoscopy, an RF current is applied to. Water vapour is delivered through a retractable vapor needle via emitter holes in the transurethral device. This is done in 9-second bursts to the transition zone of the prostate, where, via convection, it diffuses evenly throughout the target tissue. The depth of the needle penetrating is approximately 10 mm.
  Upon contact with body-temperature tissue, the water vapour then condenses. This phase shift to a liquid state dispenses concentrated energy onto the cell membranes of the target tissue, triggering instant cell necrosis. Overlapping injection sites can be established with repeated applications in order to fully target areas of hypertrophy. Saline flush irrigation is used to both cool the urethra and to promote visualization.
  At the end of the procedure Urethral catheter is fixed for 1-3 days.

SUMMARY:
new treatment modality for BPH , less invasive and more effective.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a common urological condition characterized by progressive increase in the size of the prostate gland. It is a disease of ageing, affecting 40% of men in their 50s and 90% of men over 90 years causing bladder outflow obstruction (BOO), which results in lower urinary tract symptoms (LUTS) which have a significant impact on quality of life (QoL).

The current management for LUTS caused by BOO secondary to BPH includes conservative approaches (watchful waiting and lifestyle modifications), pharmacotherapy and surgical intervention.

The Surgical interventions include open surgery (suprapubic and perineal approaches),transurethral resection of the prostate (TURP) which was a revolutionary step in the management of BPH, and was considered the first minimally invasive treatment for prostate enlargement and With the improvement of endoscopes, development and incorporation of new technologies into the medical field, minimally invasive procedures have been more and more introduced as surgical options to treat BPH .

Minimally invasive procedures include water vapor thermal therapy (REZUM), trans urethral needle ablation, trans urethral microwave thermotherapy, prostate urethral lift and prostate artery embolization.

REZUM (water vapor thermal therapy) is considered one of the advanced minimal invasive procedure that uses the principles of convective heat transfer that exploits the thermodynamic properties of water to remove the excess prostate tissue that is pressing on the urethra.

The therapy is targeted to a defined area because steam will travel only between cells until it encounters natural collagen barriers or the prostate capsule itself.

After the REZUM procedure, the body creates an inflammatory response, which takes two to four months to completely resolve. Initially, there will be swelling in the prostate, which can cause restriction of flow and cause more difficulty and frequency of urination.

In general, after the procedure symptoms will get worse before they get better and improved.

Erections are not affected by the REZUM procedure and there is 1% to 2% chance of retrograde ejaculation and his is a significantly lower percentage than in other prostate procedures.

Advantages of REZUM:

* Can be performed under sedation only
* Day case procedure
* Strong short-term safety profile
* No reports of de novo sexual dysfunction
* Suitable for patients with an obstructing median lobe
* Short procedure time
* Good improvement in subjective and objective outcome measures: IPSS, QoL, Qmax and PVR
* Cost effective

Disadvantages of REZUM:

* Limited long-term data available
* Not suitable for patients with history of recurrent urinary tract infections
* Not suitable for large prostate size (>120 cc)
* Not suitable for patients if prior invasive procedure for treatment of prostate or prior radiation on prostate
* >50% patients require catheter post procedure

ELIGIBILITY:
Inclusion Criteria:

* any patient diagnosed with BPH

Exclusion Criteria:

* PATIENT REFUSING TO PARTICIPITATE

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of the IPSS | 1 month after treatment
  to assess the success of treatment ,pre-operative and postoperative questionnaire will be done
duration of the operation | intra-operative
  minutes or hours needed for the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Gadalmoulah, phd, Study Director — professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang SJ, Qian HN, Zhao Y, Sun K, Wang HQ, Liang GQ, Li FH, Li Z. Relationship between age and prostate size. Asian J Androl. 2013 Jan;15(1):116-20. doi: 10.1038/aja.2012.127. Epub 2012 Dec 10. PMID 23223031
- [Background] Vuichoud C, Loughlin KR. Benign prostatic hyperplasia: epidemiology, economics and evaluation. Can J Urol. 2015 Oct;22 Suppl 1:1-6. PMID 26497338
- [Background] Kim EH, Larson JA, Andriole GL. Management of Benign Prostatic Hyperplasia. Annu Rev Med. 2016;67:137-51. doi: 10.1146/annurev-med-063014-123902. Epub 2015 Sep 2. PMID 26331999
- [Background] Magistro G, Chapple CR, Elhilali M, Gilling P, McVary KT, Roehrborn CG, Stief CG, Woo HH, Gratzke C. Emerging Minimally Invasive Treatment Options for Male Lower Urinary Tract Symptoms. Eur Urol. 2017 Dec;72(6):986-997. doi: 10.1016/j.eururo.2017.07.005. Epub 2017 Jul 19. PMID 28734706
- [Background] Garden EB, Shukla D, Ravivarapu KT, Kaplan SA, Reddy AK, Small AC, Palese MA. Rezum therapy for patients with large prostates (>/= 80 g): initial clinical experience and postoperative outcomes. World J Urol. 2021 Aug;39(8):3041-3048. doi: 10.1007/s00345-020-03548-7. Epub 2021 Jan 3. PMID 33392646
- [Background] Elterman D, Shepherd S, Saadat SH, Alshak MN, Bhojani N, Zorn KC, Rijo E, Misrai V, Lajkosz K, Chughtai B. Prostatic urethral lift (UroLift) versus convective water vapor ablation (Rezum) for minimally invasive treatment of BPH: a comparison of improvements and durability in 3-year clinical outcomes. Can J Urol. 2021 Oct;28(5):10824-10833. PMID 34657655